CLINICAL TRIAL: NCT01264016
Title: Performance of the TATSU/Tradewind Blood Glucose Monitoring System
Brief Title: Performance of a New Glucose Meter System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ascensia Diabetes Care (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CTD-2010-004-01
Record Dates: First submitted 2010-12-18; First posted 2010-12-21 (Estimated); Results first posted 2012-05-01 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-01

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intended Users of the Monitoring System (Experimental): Untrained subjects with diabetes use an investigational blood glucose monitoring system.
  Interventions: Device: Investigational Blood Glucose Monitoring System

INTERVENTIONS:
Device: Investigational Blood Glucose Monitoring System — Untrained subjects with diabetes performed Blood Glucose (BG) tests with subject's capillary fingerstick using the investigational Tradewind meter and investigational sensor. Study staff tested subject venous blood. All BG Results were compared to a reference laboratory glucose method. Subjects' success at performing basic tasks using only the User Guide were rated by study staff.

SUMMARY:
The purpose of this study is to evaluate the performance and acceptability of a new blood glucose monitoring system, which includes meter and sensor strip.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or 2 diabetes
* Age 18 years or older
* Routinely performs blood glucose self testing at home, at least once per day
* Able to speak, read, and understand English.
* Is willing to complete all study procedures

Exclusion Criteria:

* Currently pregnant
* Hemophilia or any other bleeding disorder
* Taking prescription anticoagulants or has clotting problems that may prolong bleeding. Taking aspirin daily is not excluded
* Subject employee of competitive medical device company
* Cognitive disorder or other condition, which in the opinion of the investigator, would put the person at risk or seriously compromise the integrity of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2010-11; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Bailey, MD, Principal Investigator — AMCR Institute
Locations (1):
- AMCR Institute, Escondido, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intended Users of the Monitoring System
Started | 96
Completed | 94
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Felt faint at sight of blood | 1

BASELINE CHARACTERISTICS:
Groups:
- Intended Users of the Monitoring System: Untrained subjects with diabetes use an investigational blood glucose monitoring system. One subject withdrew voluntarily; one subject was withdrawn. One subject hematocrit measurement was missing so subject data was not evaluable.
Arm/Group | Intended Users of the Monitoring System
Number analyzed (Participants) | 93
Age, Continuous [Mean (Full Range); unit: years]
  Mean age (range of ages) | 37.8 [18 to 73]
Sex: Female, Male [Count of Participants; unit: Participants] — 94 subjects completed study; 93 subjects had evaluable blood glucose data as described in outcome measure results
  Participants
    Female | 47
    Male | 46
Region of Enrollment [Number; unit: participants] — One subject withdrew voluntarily; one subject was withdrawn. 94 subjects completed the study.
  participants
    United States | 93

OUTCOME MEASURES:

1. Primary Outcome: Percent of Capillary Blood Glucose (BG) Results Within +/- 5 to 20mg/dL (<75 mg/dL) or Within +/- 5% to 20% (>=75 mg/dL) of Laboratory Glucose Method
Description: Subjects with diabetes used an investigational blood glucose monitoring system (BGMS) with subject capillary blood. BGM results were compared to a reference lab glucose method - Yellow Springs Instrument (YSI) Analyzer. BG results were used to calculate the number of BG results within +/- 5 to 20 mg/dL (for reference BG results <75mg/dL) or +/- 5 to 20% (for reference BG results >=75mg/dL) of the reference method results.
Time Frame: 2 hours
Population: One subject did not complete capillary blood testing (low blood sugar) and one subject hematocrit measurement was missing. These subjects' blood test data was not evaluable. Since the remaining 92 subjects tested 2 test strip lots on the BGM system, 2x92(184) tests results were possible.
Measure: Number; unit: percentage of BG Results
Units Other Than Participants: blood glucose test results
Arm/Group | Intended Users of the Monitoring System
Number analyzed (Participants) | 92
Number analyzed (blood glucose test results) | 184
percentage of BG Results
  % within 20mg/dL (<75mg/dL BG) | 100.0
  % within 20mg/dL (>=75mg/dL BG) | 100.0
  % within 15mg/dL (<75 mg/dL BG) | 100.0
  % within 15mg/dL (>=75 mg/dL BG) | 100.0
  % within 10mg/dL (<75 mg/dL BG) | 100.0
  % within 10mg/dL (>=75 mg/dL BG) | 98.2
  % within 5mg/dL (<75 mg/dL BG) | 80.0
  % within 5mg/dL (>=75 mg/dL BG) | 75.0

2. Primary Outcome: Percent of Venous Blood Glucose (BG) Results Within +/- 5 to 20 mg/dL (<75 mg/dL) or Within +/- 5% to 20% (>=75 mg/dL) of Laboratory Glucose Method
Description: Healthcare professionals (study staff) used an investigational blood glucose monitoring system (BGMS) with subject venous blood. BGM results were compared to a reference lab glucose method - Yellow Springs Instrument (YSI) Analyzer. BG results were used to calculate the number of BG results within +/- 5 to 20 mg/dL (for reference BG results <75mg/dL) or +/- 5% to 20% (for reference BG results >=75mg/dL) of the reference method results.
Time Frame: 2 hours
Population: One subject's hematocrit measurement was missing, so this subject's blood test data was not evaluable. Since study staff tested each subject's venous blood using 2 lots of test strips, 2x93(or 186) test results were possible.
Measure: Number; unit: percentage of venous bg results
Units Other Than Participants: venous blood glucose test results
Groups:
- Study Staff Test Subject Venous Blood: Healthcare professionals (study staff) used an investigational blood glucose monitoring system (BGMS) with subject venous blood.
Arm/Group | Study Staff Test Subject Venous Blood
Number analyzed (Participants) | 93
Number analyzed (venous blood glucose test results) | 186
percentage of venous bg results
  % within 20mg/dL (<75mg/dL bg) | 100.0
  % within 20mg/dL (>=75mg/dL bg) | 100.0
  % within 15mg/dL (<75mg/dL bg) | 100.0
  % within 15mg/dL (>=75mg/dL bg) | 100.0
  % within 10mg/dL (<75mg/dL bg) | 100.0
  % within 10mg/dL (>=75mg/dL bg) | 98.8
  % within 5mg/dL (<75mg/dL bg) | 87.5
  % within 5mg/dL (>=75mg/dL bg) | 82.9

3. Secondary Outcome: Number of Subjects Rated as<=3 Performing Basic Meter Tasks (Labeling Comprehension)
Description: Subjects reviewed the instructions for use (User Guide and Quick Reference Guide) to learn to use the system. Study staff then observed and rated the subjects (1 to 4) on their success at performing five tasks. Scale: 1.Success in performing tasks correctly without assistance. 2.Successful with additional review of User Guide. 3.Successful with additional review and study staff assist similar to review of a specific function during a Customer Service call. 4.Subject did not perform task correctly and study staff intervention was required.
Time Frame: 2 hours
Population: Per protocol
Measure: Number; unit: participants
Arm/Group | Intended Users of the Monitoring System
Number analyzed (Participants) | 94
participants
  Turn meter on/off | 94
  Date and Time Set on Meter | 92
  Normal Control Testing | 94
  Subject blood testing | 94
  Understand underfill icon/ability to apply more bl | 94

ADVERSE EVENTS:
Time Frame: Each subject participated for approximately 2 hours.
Arm/Group | Intended Users of the Monitoring System
Serious Adverse Events (participants affected / at risk) | 0/96
Other Adverse Events (participants affected / at risk) | 13/96
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intended Users of the Monitoring System (N=96)
Hypoglycemia (Endocrine disorders) | 13 (13) — Since the subjects were people with diabetes, these hypoglycemia adverse events were anticipated and not related to the device. Also, all adverse events were mild.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days